CLINICAL TRIAL: NCT05211986
Title: An Open-label Dose Escalation Study to Assess the Safety and Tolerability of IMM01-STEM in Participants With Muscle Atrophy Related to Knee Osteoarthritis
Brief Title: Safety and Tolerability of IMM01-STEM in Patients With Muscle Atrophy Related to Knee Osteoarthritis.
Acronym: STEM-MYO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STEM-MYO
Record Dates: First submitted 2021-11-29; First posted 2022-01-27 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: 4 dose cohorts: Cohort A, IMM01-STEM 225μg; Cohort B, IMM01-STEM 450 μg; and Cohort C, IMM01-STEM 900 μg; Cohort D, IMM01-STEM 2000μg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Active Comparator): Participants will receive twice weekly intramuscular (im) administration of IMM01-STEM for 4 weeks with a dose of 225μg.
  Interventions: Drug: IMM01-STEM
- Cohort B (Active Comparator): Participants will receive twice weekly intramuscular (im) administration of IMM01-STEM for 4 weeks with a dose of 450μg.
  Interventions: Drug: IMM01-STEM
- Cohort C (Active Comparator): Participants will receive twice weekly intramuscular (im) administration of IMM01-STEM for 4 weeks with a dose of 900μg.
  Interventions: Drug: IMM01-STEM
- Cohort D (Active Comparator): Participants will receive twice weekly intramuscular (im) administration of IMM01-STEM for 4 weeks with a dose of 2000μg.
  Interventions: Drug: IMM01-STEM

INTERVENTIONS:
Drug: IMM01-STEM — IMM01-STEM is a secretome product derived from partially differentiated pluripotent stem cells that contains regenerative molecules.

SUMMARY:
An open-label dose escalation study to assess the safety and tolerability of IMM01-STEM in participants with muscle atrophy related to knee osteoarthritis

DETAILED DESCRIPTION:
This will be an open-label, dose escalation study to assess the safety and tolerability of IMM01-STEM, a secretome product derived from partially differentiated pluripotent stem cells that contains regenerative molecules, in participants with muscle atrophy related to knee osteoarthritis (KOA).

Up to 18 participants will receive twice weekly intramuscular administration of IMM01-STEM for 4 weeks in up to 4 dose cohorts: Cohort A, IMM01-STEM 225μg; Cohort B, IMM01-STEM 450 μg; and Cohort C, IMM01-STEM 900 μg; Cohort D, IMM01-STEM 2000 μg.

Study participants will sign a written Informed Consent Form (ICF) prior to the conduct of any study related procedures. A study participant who provides written informed consent will be screened within 28 days prior to treatment. Screening assessments will be conducted, after which the study participants' eligibility will be determined on the basis of the inclusion and exclusion criteria.

Eligible participants will be enrolled and undergo Baseline assessments on Day 1. Patients will receive IMM01-STEM twice a week for 4 weeks, for a total of 8 injections. Site staff will administer study medication by im injection using a small-gauge needle (eg, 24 or 26 Ga) at all scheduled visits. After each administration of study medication, participants will be observed for 3 hours to monitor for injection-related reactions and other early onset treatment-related adverse events (AEs), in particular for the presence of allergic reactions. After Visit 2 and 3, there will be follow-up phone contact 6 to 8 hours later the same day and once the day following each injection.

After their last injection, participants will enter a Safety Follow-Up (SFU) period, with clinic visits 3 days after their last injection and then monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Has moderate KOA (defined as Kellgren-Lawrence [KL] grade 2 to 3) on affected limb
* Has quadriceps weakness (<7.5N/kg)
* Can ambulate >50 feet unassisted
* This criteria deleted with protocol amendment 6
* Has a body mass index (BMI) of <40kg/m2
* A male must agree to use contraception during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
* A female is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP). OR
  2. A WOCBP who agrees to follow the protocol's contraceptive guidance during the treatment period and for at least 3 months after the last dose of study treatment.
* Female has a negative pregnancy test result at screening and prior to investigational medicinal product (IMP) administration
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
* Willing and able to comply with all study requirements, according to the judgment of the Investigator
* Has discontinued systemic oral or intravenous steroid use for 6 months prior to Screening
* Has vital sign measurements within the following ranges at Baseline (predose at Visit 2): heart rate >50 and <100 bpm, systolic blood pressure >100 and <170 mmHg, diastolic blood pressure >50 and <90 mmHg, and blood oxygenation (by pulse-oximetry) >95%
* Participant has undergone and failed at least 1 3-month or longer treatment regimen (ie, activity modification, weight loss, physical therapy, anti-inflammatory medications, or injection therapy) within a 2-year period prior to the Screening visit.
* Study participant is able to speak, read, and understand English, in order to understand the nature of this study.

Exclusion Criteria:

* Severe KOA (defined as KL grade >3) on contralateral limb
* Has had prior total knee arthroplasty
* Has a known hypersensitivity to any components of the study medication or comparative drugs (and/or an investigational device) as stated in this protocol
* Has current or past history of malignancy (5y) excluding nonmelanoma skin cancer
* Has neurological, vascular, or cardiac condition that limit function, or, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Has uncontrolled comorbidities including diabetes (hemoglobin A1c level >7.0%), Hypertension (resting heart rate >100 bpm, systolic blood pressure >170 mmHg, or diastolic blood pressure >90 mmHg), cardiovascular disease, asthma, or COPD.
* Is known positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb) or human immunodeficiency virus-1/2 antibody (HIV-1/2Ab). Patients with a negative RNA test for HCV are acceptable.
* Is taking a prohibited medication or has taken a prohibited medication (narcotic pain medication, local anti-inflammatory, other investigational drugs)
* Participant has had a change in medication to manage comorbid condition(s) (including diabestes, hypertension, asthma, and cardiovascular disease) within 1 month of the Screening visit.
* Participant received intra-articular cortisone or viscosupplementation product(eg, Synvisc®) injections within 3 months prior to the first dose of IMP.
* Has had administration of a live, attenuated vaccine within 28 days of starting study treatment or anticipation that such vaccine will be required during the study Prior/concurrent clinical study experience
* Has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* This criteria was deleted with protocol amendment 6
* This criteria was deleted with protocol amendment 6
* This criteria was deleted with protocol amendment 6
* Has current or past history (10y) of smoking
* Has a history of chronic alcohol or drug abuse within the previous 3 months
* Participant is currently using a systemic oral or intravenous steroid regimen (eg, for asthma or other chronic respiratory condition) or brief course of systemic pulse steroid administration (eg, for flare up of nonarthritic condition or COVID-19).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of IMMUNA(IMM01-STEM) treatment in study participants with muscle atrophy related to KOA | Day 0 to Day 28
  Determined by the incidence and severity of dose-limiting toxicities (DLTs) and the incidence of treatment-emergent adverse events (TEAEs). Adverse events (AE) are classified based on Common Terminology Criteria for Adverse Events (CTCAE) as follows: Grade 0 = no adverse events, Grade 1= mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = fatal adverse events. A DLT is defined as any AE related to IMM01-STEM of a Grade 2 unresolved within 48 hours post-injection, or any Grade 3, 4, or 5 related to IMM01-STEM during any time of treatment or during the 48-hour, acute/subacute observation period.

SECONDARY OUTCOMES:
Safety and tolerability of IMMUNA(IMM01-STEM) after 4 weeks of treatment in study participants with muscle atrophy related to KOA | Day 28
  Determined by incidence, type and severity of adverse events graded according to CTCAE v5.0 and CRS revised grading system and defined by clinical relevant findings at day 28 post-treatment, or worsening of previous findings from baseline at day 28 post treatment in: self-reporting, physical examination, vital signs (body temperature, body weight, blood pressure, and heart rate), laboratory data (hematology, clinical chemistry, and urinalysis).
Functionality of the knee joint after 4 weeks of treatment with IMMUNA(IMM01-STEM) in study participants with muscle atrophy related to KOA | Day 28
  Determined by evaluation of participants with changes from baseline at day 28 post treatment in: muscle strength (measured by isometric knee extensor torque), physical function (measured by the 6-minute walk test), Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lane, PhD, Study Director — Chief Science Officer at Immunis, Inc.
Locations (2):
- United States (2):
  - Orthopaedic Specialty Institute, Irvine, California
  - University of California, Irvine - Alpha Stem Cell Clinic, Orange, California

IPD SHARING:
Plan to Share IPD: No